CLINICAL TRIAL: NCT05168475
Title: Biologics in Refractory Vasculitis (BIOVAS): A Pragmatic, Randomised, Double-blind, Placebo-controlled, Modified-crossover Trial of Biologic Therapy for Refractory Primary Non-ANCA Associated Vasculitis in Adults and Children
Brief Title: Biologics in Refractory Vasculitis: A Trial of Biologic Therapy for Refractory Primary Non-ANCA Associated Vasculitis
Acronym: BIOVAS
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: NIHR withdrawal of funding
Sponsor: Cambridge University Hospitals NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, David Jayne, Honorary Consultant Physician, Cambridge University Hospitals NHS Foundation Trust
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: BIOVAS
Record Dates: First submitted 2021-12-09; First posted 2021-12-23 (Actual); Results first posted 2025-06-17 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-05

CONDITIONS: Giant Cell Arteritis; Takayasu Arteritis; Cogan Syndrome; Relapsing Polychondritis; Cryoglobulinemic Vasculitis; IgA Vasculitis; Polyarteritis Nodosa; Cutaneous Polyarteritis Nodosa; Primary Angiitis of Central Nervous System
Keywords: vasculitis
MeSH Terms: conditions — Giant Cell Arteritis; Takayasu Arteritis; Cogan Syndrome; Polychondritis, Relapsing; Cryoglobulinemia, Familial Mixed; IgA Vasculitis; Polyarteritis Nodosa; Vasculitis | interventions — Rituximab; Infliximab; tocilizumab

STUDY DESIGN:
Intervention Model Description: Modified-crossover; participants are randomised to a fixed sequence of 4 trial IMPs. Each sequence will consist of 3 active IMP treatments and a placebo. The order of the IMPs in each sequence will be randomly allocated (e.g. RTX-INF-TCZ-PBO or INF-PBO-RTX-TCZ) from a list of 24 permutations. Further, the placebo in each sequence will be randomly allocated to mirror the drug administration schedule of 1 of the active IMPs in order to maintain the blind resulting in 72 different possible permutations
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Double-blind to patient and trial team. Pharmacy and central coordinator unblinded to minimise risk
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Rituximab (Active Comparator): Rituximab 1g IV on Days 1, 15 (+/-3d), 180 (+/-14d), 360 (+/-14d) and 540 (+/-14d). (Children, 750mg/m2/dose, maximum 1 g per dose).
  Interventions: Biological: Infliximab; Biological: Tocilizumab
- Infliximab (Active Comparator): Infliximab 5mg/kg IV on days 1, 15(+/- 3d), 43 (+/-3d), 70 (+/-3d) then every 56 days (+/-14d) thereafter.
  Interventions: Biological: Rituximab; Biological: Tocilizumab
- Tocilizumab (Active Comparator): Tocilizumab 8mg/kg IV (maximum 800mg) every 30 days (+/- 7d); 10 mg/kg (maximum 800 mg) for children < 30 kg.
  Interventions: Biological: Rituximab; Biological: Infliximab
- Placebo (Placebo Comparator): Placebo may be to one of the active biologics (ie placebo to Rituximab, Placebo to Infliximab, placebo to Tocilizumab). Only 1 placebo is in a randomised sequence of interventions.
  Interventions: Biological: Rituximab; Biological: Infliximab; Biological: Tocilizumab

INTERVENTIONS:
Biological: Rituximab — Hospital stock of rituximab used as intervention; biosimilars are allowed
  Arms: Infliximab; Placebo; Tocilizumab
Biological: Infliximab — Hospital stock of infliximab is used in the trial; biosimilars are allowed
  Arms: Placebo; Rituximab; Tocilizumab
Biological: Tocilizumab — Hospital-supplied stock.
  Arms: Infliximab; Placebo; Rituximab

SUMMARY:
Vasculitis occur when the body's immune system, rather than protecting the body, attacks blood vessels, causing injury to the vessel and the part of the body it supplies with blood. Vasculitis is rare, and there are a number of different types, which can affect both adults and children. We treat vasculitis with steroids and drugs aiming to damp down the activity of the immune system, but they often cause side effects. Some patients do not improve with this treatment, or cannot tolerate it and their vasculitis worsens; this is known as refractory vasculitis. Patients with refractory vasculitis are at high risk of health complications from the disease and its therapy and are in need of newer more effective treatments with fewer side effects.

Biologics are drugs which are designed to precisely target parts of the immune system and may have fewer side effects. Biologics have been used for several years to treat vasculitis, particularly anti-neutrophil cytoplasmic antibody (ANCA)-associated vasculitis or AAV. However, for many of the rarer types of vasculitis, and especially those vasculitis disease types that are not ANCA-associated, there is little information to support use of biologic therapies as effective treatments.

The purpose of this trial is to find out whether biologics are effective and represent value for money for participants with refractory vasculitis. The trial will include patients with Non-ANCA-associated vasculitis (NAAV)

DETAILED DESCRIPTION:
The trial is a multi-centre, randomised, double-blind, placebo-controlled, modified-crossover design which will investigate three biologics, Infliximab, Rituximab, Tocilizumab, and placebos to each, in the treatment of refractory non-ANCA-associated Vasculitis (NAAV) in adults and children. Eligible patients are randomised to a sequence of up to 4 interventions (comprising 3 biologics and 1 placebo to one of the three biologics being studied). Patients remain on first intervention in their randomised sequence for up to 2 years, or until they are deemed to fail treatment or experience a severe disease relapse, at which point they will be switched to the next intervention in their randomised sequence. When a patient switches to the next intervention in their randomised sequence, they will again remain on treatment either until the end of treatment period or until they fail treatment or experience a severe disease relapse. Patients remain on the treatment period for a maximum of 2 years, or until they have failed/experienced severe relapses on every treatment in their randomised sequence, whichever is sooner. Patients will be assessed for disease activity and relapse every 120 days up to D720.

ELIGIBILITY:
Inclusion Criteria:

1. Aged at least 5 years
2. Have given, or their parent/ legal guardian aged ≥ 16 years old has given, written informed consent
3. Diagnosis of NAAV (Appendix 4)
4. Refractory disease defined by:

   * Active disease, BVASv3-BIOVAS/ PVAS with ≥ 1 severe (new/worse) or ≥ 3 non-severe (new/worse) items despite 12 weeks of conventional therapy prior to screening visit OR
   * Inability to reduce prednisolone below 15mg/day or (0.2mg/kg/day in case of children) without relapse in the 12 weeks prior to screening visit

Exclusion Criteria:

1. Previous treatment failure/contraindication to ≥ 2 active trial IMPs
2. Increase in the dose or frequency of background immunosuppressive (e.g. methotrexate) or anti-cytokine therapy within 30 days of screening visit
3. Use of intravenous immunoglobulins within 30 days, or cyclophosphamide or lymphocyte depleting biologic (e.g. rituximab) within 6 months of screening visit
4. Concomitant use of any biologic and/or anti-TNF agent other than the trial IMPs during the trial period
5. Have an active systemic bacterial, viral or fungal infection, or tuberculosis
6. Hepatitis B (HB) core antibody (Ab) or HB surface antigen positive or hepatitis C antibody positive or human immunodeficiency virus (HIV) antibody test positive
7. History of malignancy within five years prior to screening visit or any evidence of persistent malignancy, except fully excised basal cell or squamous cell carcinomas of the skin, or cervical carcinoma in situ which has been treated or excised in a curative procedure
8. Pregnant or breastfeeding, or inability/unwillingness to use a highly effective method of contraceptive if a woman of childbearing potential (WOCBP;see section 11.9)
9. Severe disease, which in the opinion of the physician prevents randomisation to placebo
10. Recent or upcoming major surgery within 45 days of screening visit
11. Leukocyte count < 3.5 x 109 cells/l, platelet count < 100 x 109 cells/l, neutrophil count of < 2 x 109 cells/l
12. ALT or ALP > 3 times the upper limit of normal
13. Symptomatic congestive heart failure (NYHA class III/IV) requiring prescription medication within 90 days of screening visit
14. Demyelinating disorders
15. History or presence of any medical condition or disease which, in the opinion of the Investigator, may place the participant at unacceptable risk because of trial participation
16. Administration of live or live attenuated vaccines within 45 days of screening
17. Have received an investigational medicinal product (IMP) within 5 half-lives or 30 days prior to screening
18. Diagnosis of adenosine deaminase type 2 (DADA2)
19. Hypersensitivity to the active IMP substance or to any of the formulation excipients

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2021-07-14 (Actual); Primary Completion 2023-11-29 (Actual); Study Completion 2023-11-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Jayne, Principal Investigator — Cambridge University Hospitals NHS Foundation Trust/University of Cambridge
Locations (5):
- United Kingdom (5):
  - Cambridge University Hospitals NHS Foundation Trust, Cambridge
  - Glasgow Royal Infirmary, Glasgow
  - Great Ormond Street Hospital NHS Foundation Trust, London
  - Guy's and St Thomas, London
  - East Kent Hospitals, Margate

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 4 participants were excluded as they did not meet the inclusion criteria
Groups:
- All Participants: Including all randomisation assignments: Infliximab, Rituximab, Tocilizumab and Placebo
Period: Period 1
Arm/Group | All Participants
Started | 20
Infliximab (Infliximab assignment) | 7
Rituximab (Rituximab assignment) | 7
Tocilizumab (Tocilizumab assignment) | 3
Placebo (Placebo assignment) | 1
Not Randomised | 2
Completed | 15
Not Completed | 5
Not completed — Protocol Violation | 1
Not completed — IMP shortage | 2
Not completed — Not randomised | 2
Period: Period 2
Arm/Group | All Participants
Started | 10 (Between period 1 and 2: death n=1, completion n=1, non-compliance n=1, withdrawal of funds n=5)
Infliximab (Infliximab assignment) | 4
Rituximab (Rituximab assignment) | 2
Tocilizumab (Tocilizumab assignment) | 4
Placebo (Placebo assignment) | 0
Completed | 9
Not Completed | 1
Not completed — IMP shortage | 1
Period: Period 3
Arm/Group | All Participants
Started | 1 (Between period 2 and 3: Consent withdrawn n=1, completion n=1, Funds withdrawn n=6, Uncontrolled disease n=1,)
Infliximab (Infliximab assignment) | 1
Rituximab (Rituximab assignment) | 0
Tocilizumab (Tocilizumab assignment) | 0
Placebo (Placebo assignment) | 0
Completed | 0
Not Completed | 1
Period: Period 4
Arm/Group | All Participants
Started (Between periods Withdrawn n=1) | 0
Completed | 0
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Rituximab | Infliximab | Tocilizumab | Placebo | Total
Number analyzed (Participants) | 7 | 7 | 3 | 1 | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 0 | 0 | 0 | 1
  Between 18 and 65 years | 4 | 5 | 2 | 1 | 12
  >=65 years | 2 | 2 | 1 | 0 | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.57 (25.55) | 48.57 (14.41) | 54.67 (21.2) | 58 (0) | 49.33 (19.22)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 6 | 2 | 1 | 15
  Male | 1 | 1 | 1 | 0 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 7 | 7 | 3 | 1 | 18
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United Kingdom | 7 | 7 | 3 | 1 | 18
Disease group [Count of Participants; unit: Participants]
  Giant Cell Arteritis | 1 | 1 | 1 | 0 | 3
  Takayasu's Arteritis | 1 | 0 | 0 | 0 | 1
  Polyarteritis Nodosa | 1 | 0 | 1 | 0 | 2
  Relapsing Polychondritis | 2 | 3 | 0 | 0 | 5
  IgA vasculitis | 1 | 3 | 1 | 1 | 6
  Cogan's syndrome | 1 | 0 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Treatment Failure
Description: Primary treatment failure is progressive disease (defined by appearance of ≥1 new/worse severe or ≥3 new/worse non-severe items) on Birmingham vasculitis activity score (BVAS) v3 modified for BIOVAS trial (BVASv3-BIOVAS) or paediatric vasculitis activity score (PVAS) within 120 days from the time of IMP commencement; or failure to achieve clinical response (see definitions below) by 120 days from the time of IMP commencement. In such cases, TTF will be recorded as zero. We report this as number of events that occurred. As arms reached the number of events to define a median, we are reporting it as number of events.
Time Frame: up to 720 days
Measure: Number; unit: treatment failures
Arm/Group | Infliximab | Rituximab | Tocilizumab | Placebo
Number analyzed (Participants) | 12 | 9 | 7 | 1
treatment failures | 5 | 3 | 1 | 0

2. Secondary Outcome: Patients Achieving Response at the 120 Day Timepoint Following Commencement of IMP
Description: Proportion of participants achieving response at the 120 day evaluation time point after the start of each IMP.
  The response status is defined by a BVAS v3-BIOVAS/ PVAS of ≤ one non-severe (no new/worse) item, prednisolone dose ≤ 50% of the dose at the start of the IMP treatment and ≤ 10mg/day (0.2 mg/kg/day for children, whichever is lower) and an ESR < 30mm/hr or CRP <10 mg/L
Time Frame: 120 days
Measure: Count of Participants; unit: Participants
Arm/Group | Infliximab | Rituximab | Tocilizumab | Placebo
Number analyzed (Participants) | 12 | 9 | 7 | 1
Participants | 1 | 5 | 3 | 1

3. Secondary Outcome: Patients Achieving Response at Any 120 Day Timepoint
Description: Proportion of participants achieving response at every 120 day evaluation time point defined by a BVAS v3-BIOVAS/ PVAS of ≤ 1 non-severe (no new/worse) item, prednisolone dose ≤ 50% of the dose at the start of the IMP treatment and ≤ 10mg/day (0.2 mg/kg/day for children, whichever is lower) and an ESR < 30mm/hr or CRP <10 mg/L
Time Frame: up to 720 days
Measure: Number; unit: Number of responders
Arm/Group | Infliximab | Rituximab | Tocilizumab | Placebo
Number analyzed (Participants) | 12 | 9 | 7 | 1
Number of responders
  Day 240 | 6 | 4 | 2 | 1
  Day 360 | 3 | 4 | 2 | 1
  Day 480 | 2 | 1 | 1 | 1
  Day 600 | 1 | 1 | 1 | 1
  Day 720 | 0 | 1 | 0 | 1

4. Secondary Outcome: Increase in Disease Related Damage Measured by Vasculitis Damage Index/Paediatric Vasculitis Damage Index (VDI/PVDI) From Start to End of an IMP Treatment
Description: VDI/PVDI scores are collected from 11 different disease categories with each positive item scoring one mark. VDI/PVDI scores can either increase or stay the same at each measurement. All damage scores are carried forward to the next assessment. The minimum score is zero and the maximum score is 63. A low score indicates less damage and therefore a better outcome. A higher score indicates more damage and a worse outcome.
  Due to the study design, participants were kept on each intervention until treatment failure and then moved to the next in their allocated sequence. Secondary outcome data were collected from the start of the first treatment without restarting collection at each crossover. Therefore, results are presented by treatment sequence. The number of participants analysed includes all participants who received the given intervention at any time during the study.
Time Frame: VDI/PVDI scores were collected every 120 days at each scheduled visit in the trial until the last assessment at day 720 at the end of trial. 120 days, 240 days, 360 days, 480 days, 600 days and 720 days
Population: Number analysed differs in each row depending on time in study for each participant.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Infliximab | Rituximab | Tocilizumab | Placebo
Number analyzed (Participants) | 12 | 9 | 7 | 1
score on a scale
  Baseline: number analyzed (Participants) | 6 | 9 | 7 | 1
  Baseline | 1 [0.25 to 1.75] | 2 [1 to 3] | 1 [0.5 to 2] | 3 [3 to 3]
  Day 120: number analyzed (Participants) | 6 | 6 | 7 | 1
  Day 120 | 1 [0.25 to 3.25] | 2 [2 to 2] | 2 [1 to 2.5] | 3 [3 to 3]
  Day 240: number analyzed (Participants) | 6 | 6 | 2 | 1
  Day 240 | 1 [1 to 3.25] | 2 [1.25 to 2.75] | 1.5 [0.75 to 2.25] | 3 [3 to 3]
  Day 360: number analyzed (Participants) | 5 | 5 | 2 | 1
  Day 360 | 1.5 [0.75 to 2.5] | 3 [2 to 3] | 1.5 [0.75 to 2.25] | 3 [3 to 3]
  Day 480: number analyzed (Participants) | 3 | 3 | 1 | 1
  Day 480 | 2 [1 to 3] | 4 [3.5 to 4.5] | 3 [3 to 3] | 3 [3 to 3]
  Day 600: number analyzed (Participants) | 2 | 2 | 1 | 1
  Day 600 | 0 [0 to 0] | 3 [2.5 to 3.5] | 3 [3 to 3] | 3 [3 to 3]
  Day 720: number analyzed (Participants) | 1 | 1 | 0 | 1
  Day 720 | 0 [0 to 0] | 4 [4 to 4] |  | 3 [3 to 3]

5. Secondary Outcome: Physician's Global Assessment (PGA) (Likert Scale 0-10)
Description: Physician's global assessment at every 120 day evaluation time point from the time of IMP commencement The Physician's global assessment (PGA) is a visual analogue scale from 0-10, where 0 is no disease activity (better outcome) and 10 is maximum disease activity (worse outcome).
  PGA scores are collected every 120 days at each scheduled visit for each participant (unless a visit is unscheduled which could occur at any time in between the time points).
  Due to the study design, participants were kept on each intervention until treatment failure and then moved to the next in their allocated sequence. Secondary outcome data were collected from the start of the first treatment without restarting collection at each crossover. Therefore, results are presented by treatment sequence. The number of participants analysed includes all participants who received the given intervention at any time during the study.
Time Frame: 120 days, 240 days, 360 days, 480 days, 600 days, 720 days
Population: Number analysed differs in each row depending on time in study for each participant
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Infliximab | Rituximab | Tocilizumab | Placebo
Number analyzed (Participants) | 12 | 9 | 7 | 1
score on a scale
  Baseline: number analyzed (Participants) | 6 | 7 | 3 | 1
  Baseline | 2.5 [2 to 3] | 4 [2.5 to 4] | 4 [3.5 to 4.5] | 5 [5 to 5]
  Day 120: number analyzed (Participants) | 6 | 6 | 3 | 1
  Day 120 | 3.5 [2.25 to 4.75] | 1.5 [1 to 2] | 1 [1 to 1.5] | 2 [2 to 2]
  Day 240: number analyzed (Participants) | 6 | 6 | 2 | 1
  Day 240 | 1 [1 to 1.75] | 1 [1 to 1] | 1 [1 to 1] | 2 [2 to 2]
  Day 360: number analyzed (Participants) | 5 | 5 | 2 | 1
  Day 360 | 1.5 [1 to 2.25] | 2 [2 to 3] | 1 [1 to 1] | 1 [1 to 1]
  Day 480: number analyzed (Participants) | 3 | 3 | 1 | 1
  Day 480 | 2.5 [2.25 to 2.75] | 1 [1 to 2.5] | 1 [1 to 1] | 1 [1 to 1]
  Day 600: number analyzed (Participants) | 2 | 2 | 1 | 1
  Day 600 | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1]
  Day 720: number analyzed (Participants) | 1 | 1 | 0 | 1
  Day 720 | 0 [0 to 0] | 1 [1 to 1] |  | 1 [1 to 1]

6. Secondary Outcome: Serious Adverse Events/Adverse Events of Special Interests (SAEs/AESIs)
Description: Serious adverse events (SAEs) and adverse events of special interest (AESI) (where infection is considered an AESI)
Time Frame: up to 720 days
Measure: Number; unit: Number of Events
Arm/Group | Infliximab | Placebo | Rituximab | Tocilizumab
Number analyzed (Participants) | 12 | 1 | 9 | 7
Number of Events
  AESI | 21 | 2 | 17 | 0
  SAE | 0 | 0 | 7 | 0

ADVERSE EVENTS:
Time Frame: 24 months
Description: Only adverse events of special interest (AESIs) as described in section 12.3 will be reported from the point of informed consent until the end of participation in the trial for each participant.
  In addition to all SAEs, all infections requiring antimicrobial, antiviral or antifungal treatment are being collected as adverse events of special interest (AESIs) as part of the BIOVAS trial.
Arm/Group | Infliximab | Rituximab | Tocilizumab | Placebo
All-Cause Mortality (participants affected / at risk) | 0/12 | 1/9 | 0/7 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/12 | 3/9 | 0/7 | 0/1
Other Adverse Events (participants affected / at risk) | 7/12 | 5/9 | 0/7 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Infliximab (N=12) | Rituximab (N=9) | Tocilizumab (N=7) | Placebo (N=1)
Tonsillitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Polychondritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oral candidiasis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
vasculitis rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Septic shock (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Infliximab (N=12) | Rituximab (N=9) | Tocilizumab (N=7) | Placebo (N=1)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Covid-19 (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
E.Coli Urinary Tract Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ear Infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Labyrinthitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Localised infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Oral candidiasis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oral Herpes (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oral infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Paronychia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pelvic Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pseudomonas infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory Tract Infection (Infections and infestations) | 4 (4) | 3 (3) | 0 (0) | 1 (1)
Skin infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
staphylococcal skin infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
systemic infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tonsillitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 3 (3) | 4 (4) | 0 (0) | 0 (0)
vulvovaginal candidiasis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
The recruitment period was planned to be 29 months, however study activities were halted after 20 months due to funding being withdrawn.

18 participants were randomised rather than the intended sample size of 140. Due to the small number of participants recruited the analyses are mainly descriptive.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication or other dissemination of the Results (or any part of them) by any of the Parties shall not occur until the Lead has published the Results of the Project in the primary publication (the "Primary Publication").

DOCUMENTS (2):
  • Study Protocol (2021-11-17): https://cdn.clinicaltrials.gov/large-docs/75/NCT05168475/Prot_000.pdf
  • Statistical Analysis Plan (2024-04-19): https://cdn.clinicaltrials.gov/large-docs/75/NCT05168475/SAP_001.pdf